CLINICAL TRIAL: NCT04323579
Title: Validation of Multiparametric Models and Circulating and Imaging Biomarkers to Improve Lung Cancer EARLY Detection.
Acronym: CLEARLY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other); University of Paris 5 - Rene Descartes (Other); Maastricht University (Other); Medical University of Gdansk (Other); Erasmus Medical Center (Other); University of Wuerzburg (Other)
Responsible Party: Sponsor
Other Study IDs: 2122
Record Dates: First submitted 2019-01-10; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- prospective cohort of stage I-II lung cancer patients: A prospective cohort of stage I-II lung cancer patients (N=80) candidates to surgery at Humanitas, and 40 controls with benign nodules.
- retrospective screening cohort of 50 patients: A retrospective screening cohort of 50 patients with screened lung cancer at MUG.
- prospective screening cohort of 30 patients: A prospective screening cohort of 30 patients with screened lung cancer and 100 matched negative controls enrolled at Humanitas cohort of 1000 participants (expected annual rate 1.5%).
- retrospective screening cohort from the NELSON study: A retrospective screening cohort from the NELSON study.
- Prospective cohort of stage IV lung cancer patients: A Prospective cohort of stage IV lung cancer patients (N=30) candidate to systemic therapy.

SUMMARY:
CLEARLY will focus on validation of a multifactorial "bio-radiomic" protocol for early diagnosis of lung cancer that combines circulating biomarkers and radiomic analysis. It will (a) assess the role of molecular and cellular biomarkers (exosomes, protein signatures, circulating tumor cells - CTCs, microRNA) and radiomic signature, as complementary to assist early detection of lung cancer by low dose computed tomography-LDCT, using bioinformatics techniques; (b) assess the prognostic role of CTCs including the role of cells epithelial mesenchymal transition (EMT) and (c) standardize a method for genomic analysis of CTCs for early detection of treatment resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years old and exposure to smoking more than 30 packs-year; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%).
* Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study.
* Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.

Exclusion Criteria:

* Previous diagnosis of lung cancer.
* Positive extrapulmonary cancer history in the last 5 years (excluding in situ tumors or skin epidermoid tumor).
* Performing a chest CT scan in the last 18 months.
* Severe lung or extrapulmonary diseases that may preclude or invalidate appropriate therapy in case of diagnosis of malignant pulmonary neoplasia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population should have the following inclusion criteria: Inclusion Criteria: - Age ≥ 55 years old and exposure to smoking more than 30 packsyear; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%). - Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study. - Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the role of a bio-radiomic protocol as complementary tool to assist early detection of lung cancer by LDCT | 01 July 2018 - 01 July 2021
  CTC analysis will be performed using fresh plasma samples. Blood collection will be obtained for each lung cancer patient before and after surgery and once for controls. 45- and 16-miRNA signatures will be analyzed on plasma samples of the retrospective cohort (150 lung cancer patients and 120 matched controls). We will perform the exosome antigens analysis in the retrospective cohort. We will validate the 8-protein signature in the retrospective cohort. We will validate the radiomic signature on CT images, and further validation will be performed on CT images of the prospective cohorts collected and 70 screened individuals of the retrospective cohort. We will integrate results of biomarkers and radiomic data and will build a multiparametric risk model to improve early detection of lung cancer. The final predictive model will be then applied to the cohorts analysed and integrated with LDCT results to evaluate the improvement in diagnostic accuracy.

SECONDARY OUTCOMES:
Correlation of CTC spread to angiogenesis. | 01 July 2018 - 01 July 2021
  Number of CTC isolated with ISET technique in the prospective cohort of lung cancer patients and controls will be correlated to angiogenesis aspects of the primary tumor at CT scan, using dynamic perfusion data and quantitative and qualitative assessment of angiogenesis (surface fractal dimension and microvessel density) on hysthological examination.
Assessment of epithelial mesenchymal transition (EMT) in CTC as a hallmark of poor prognosis. | 01 July 2018 - 01 July 2021
  The presence of CTC passed through EMT will be identified using immunoistochimical specific exams. The correlation between the presence of CTCs in EMT and prognostic factors of primary tumor (disease stage, volume doubling time, etc) will show the possible prognostic role of CTC immunoistochemical analysis.
Standardise a method for genomic analysis from isolated CTCs for the early detection of resistance to treatments | 01 July 2018 - 01 July 2021
  A population of patients with advanced stage disease (stage III and IV) will be first analyzed to enrich for CTCs in the collected blood samples. This would help the initial refinement of the experimental protocol to detect CTC and analyse their mutational profile by single-cell NGS analysis. In addition, since most of these patients will undergo systemic treatment, we will setup a longitudinal study where the mutational profile of CTC will be investigated and correlated to chemotherapy response, to early identify theranostic mutations. The same refined protocol will be next validated on the prospective cohort of LDCT screened patients to further prove its validity to early detect cancer driver mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy